CLINICAL TRIAL: NCT00055328
Title: Problem-Solving Treatment for Primary Care Depression
Brief Title: Treatment for Depression in the Primary Care Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH062322 (NIH); R01MH062322 (NIH); DATR A4-GPS
Record Dates: First submitted 2003-02-25; First posted 2003-02-26 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2008-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Primary Health Care

INTERVENTIONS:
Behavioral: Problem-Solving Treatment for Primary Care

SUMMARY:
This study will compare a brief form of counseling to usual care for the treatment of minor depression in the primary care setting.

DETAILED DESCRIPTION:
Minor depression is one of the most common types of depressive disorders seen in primary care. The effectiveness and tolerability of antidepressants in patients with minor depression is unclear, and the development of alternative treatments is necessary.

In the first phase of this study, participants are observed for 4 weeks to identify those most in need of depression-specific treatment. Participants are then exposed to the Problem-Solving Treatment for Primary Care (PST-PC), a six-session behavioral treatment for depression. After 4 weeks, patients who do not respond adequately to the treatment are randomly assigned to either continued PST-PC or to usual care for 9 weeks. Participants are followed for 6 months after the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary care patient at Dartmouth-Hitchcock Medical Center (DHMC)
* Hamilton Depression Score >= 10 and minor depression at time of entry and after 4 weeks of observation

Exclusion Criteria:

* Psychosis, Obsessive Compulsive Disorder (OCD), or Post Traumatic Stress Disorder (PTSD)
* Active substance abuse
* Receiving treatment for depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-12; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States